CLINICAL TRIAL: NCT04508595
Title: The RestEaze Ambulatory Sleep Monitor for Detection of Leg Movements During Sleep in Adults and Children With a Sleep Disturbance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanzen Medical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: TM-RE1-OBS-0001
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Sleep

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: RestEaze — Wearable band to detect leg movements of sleep

SUMMARY:
This observational study will test and evaluate the RestEaze ambulatory sleep monitor for the detection and classification of leg movements during sleep (LMS) and other sleep measures.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 5 -75
* General good health and ambulatory
* Sleep complaint or other diagnosis that affects sleep (e.g. ADHD) with likely concomitant abnormal LMS requiring either HST or PSG
* Reports no significant problems sleeping in a new bed and bedroom away from home
* (If applicable) Parent or guardian available to spend the night with the child during the sleep study

Exclusion Criteria:

• Amputation that would preclude use of wrist actigraph or the RestEaze device

Ages: 5 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients presenting to sleep medicine clinic for evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-08 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-08-06 (Estimated)

PRIMARY OUTCOMES:
Algorithm | 1 year
  Development of analysis tools to validate RestEaze as a biomarker of leg movements of sleep

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Sleep Center, Milpitas, California, United States

IPD SHARING:
Plan to Share IPD: No